CLINICAL TRIAL: NCT03418389
Title: An Observational, Longitudinal Study to Evaluate and Monitor Physical Performance of Adults Treated With Asfotase Alfa for Pediatric-Onset Hypophosphatasia
Brief Title: Evaluate and Monitor Physical Performance of Adults Treated With Asfotase Alfa for Hypophosphatasia
Acronym: EmPATHY
Status: Completed | Type: Observational
Sponsor: Dr. Lothar Seefried (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Lothar Seefried, Head, Clinical Trial Unit, Orthopedic Department, Wuerzburg University Hospital
Organization: Wuerzburg University Hospital (Other)
Other Study IDs: KLH-01-2018
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric-onset Hypophosphatasia

SUMMARY:
Hypophosphatasia is a rare inherited metabolic disorder due to inactivating mutations of the ALPL-Gene. Particularly among adult patients, clinical manifestation exhibits a broad range of signs and symptoms, most commonly associated with musculoskeletal disabilities and compromised quality of life. Enzyme replacement therapy with Asfotase alfa (AA) is available and approved for patients with pediatric onset of the disease.

This single-center observational cohort study aims at collecting clinical routine data regarding the course treatment, quality of life and physical performance in patients treated with Asfotase alfa in line with the label for pediatric-onset hypophosphatasia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of enrollment
* Clinical diagnosis of pediatric-onset HPP based on low ALP (age- and sex-adjusted) and/or genetic confirmation of ALPL mutation(s), and clinical symptoms consistent with HPP
* Participant currently receiving commercial asfotase alfa treatment for HPP at the Orthopedic Institute of the Julius-Maximilians-University Würzburg, as per standard of care
* Willingness to participate in the study
* Signed informed consent

Exclusion Criteria:

* Unwillingness / anticipated inability to attend further visits
* Off-label treatment with asfotase alfa
* Current participation in an Alexion Sponsored Trial
* Experimental drug/treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of male and female HPP patients with pediatric-onset HPP currently being managed for the disease at the Orthopedic Institute of the Julius-Maximilians-University Würzburg, Germany and receiving commercial AA treatment as per the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  6 Minute Walk Test [meters]
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  Short Physical Performance Battery [points]
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  Timed Up and Go Test [seconds]
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  Handheld dynamometry [kilogram]
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  Jumping mechanography [W/kg bodyweight]
Physical Performance | 1 year of treatment compared to pre-treatment baseline
  Use of assistive devices descriptive measure
Body composition | 1 year of treatment compared to pre-treatment baseline
  Bioelectrical Impedance Analysis [proportional mass of muscle, water and fat in kg]

SECONDARY OUTCOMES:
Health related quality of life | 1 year of treatment compared to pre-treatment baseline
  Questionnaire
Bone Mineral Density | 1 year of treatment compared to pre-treatment baseline
  Dual x-ray absorptiometry (DXA)
Skeletal pathology | 1 year of treatment compared to pre-treatment baseline
  Descriptive assessment of available imaging (x-Ray, CT, MRI, histological sections)
Laboratory evaluation | 1 year of treatment compared to pre-treatment baseline
  Parathyroid hormone [PTH, pg/ml]
Laboratory evaluation | 1 year of treatment compared to pre-treatment baseline
  Serum-Calcium [mmol/l]
Laboratory evaluation | 1 year of treatment compared to pre-treatment baseline
  Serum-Phosphorus [mmol/l]
Laboratory evaluation | 1 year of treatment compared to pre-treatment baseline
  Serum-Creatinine [µmol/l], incl. calculated eGFR
Laboratory evaluation | 1 year of treatment compared to pre-treatment baseline
  Fibroblast Growth Factor 23 / FGF-23 [RU/ml]
Safety assessment | 1 year of treatment compared to pre-treatment baseline
  Injection site reactions (descriptive)
Safety assessment | 1 year of treatment compared to pre-treatment baseline
  Injection associated reactions (descriptive)
Safety assessment | 1 year of treatment compared to pre-treatment baseline
  Ectopic calcifications (descriptive)
Safety assessment | 1 year of treatment compared to pre-treatment baseline
  Adverse events (descriptive)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Seefried, MD, Principal Investigator — Wuerzburg University, Orthopedic Institute, Clinical Trial Unit
Locations (1):
- Clinical Trial Unit, Orthopedic Department, Wuerzburg University, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seefried L, Genest F, Petryk A, Veith M. Effects of asfotase alfa in adults with pediatric-onset hypophosphatasia over 24 months of treatment. Bone. 2023 Oct;175:116856. doi: 10.1016/j.bone.2023.116856. Epub 2023 Jul 20. PMID 37481150